CLINICAL TRIAL: NCT04552327
Title: Prospective, Three-armed, Randomised, Double-blind Study to Evaluate the Efficacy and Safety of the Treatment of Mild and Moderate Actinic Keratosis With a 5% Potassium Hydroxide Solution (Solcera, Medical Device) Versus Placebo and Investigator-blinded Comparison With 3% Diclofenac Gel (Solaraze, Medicinal Product) (Regulated by the Laws for Both Medical Devices and Medicinal Products)
Brief Title: 5% KOH Solution vs. Placebo and Diclofenac Gel for the Treatment of Actinic Keratosis
Acronym: KOHDIAK
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Infectopharm Arzneimittel GmbH (Industry)
Collaborators: Gesellschaft für Therapieforschung mbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KOHDIAK
Record Dates: First submitted 2020-09-03; First posted 2020-09-17 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-02

CONDITIONS: Actinic Keratosis
Keywords: Actinic Keratosis; Solcera; Prospective; Multicentric; Monitored; Efficacy; Safety; Potassium Hydroxide; Randomized; Double-Blind
MeSH Terms: conditions — Keratosis, Actinic | interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Solcera (Experimental)
  Interventions: Device: Solcera
- Placebo (Placebo Comparator)
  Interventions: Device: Placebo
- Solaraze (Active Comparator)
  Interventions: Drug: Solaraze

INTERVENTIONS:
Device: Solcera — Twice daily application for a duration of 4 weeks followed by another 4 weeks without treatment (up to 2 potential repetitions of this 8-week cycle)
  Arms: Solcera
Device: Placebo — Twice daily application for a duration of 4 weeks followed by another 4 weeks without treatment (up to 2 potential repetitions of this 8-week cycle)
  Arms: Placebo
Drug: Solaraze — Twice daily application for a duration of 60 days
  Arms: Solaraze

SUMMARY:
The KOHDIAK study is a prospective, three-armed, randomised, double-blind study to evaluate the efficacy and safety of the treatment of mild and moderate actinic keratosis with a 5% potassium hydroxide solution (Solcera, medical device) versus placebo and investigator-blinded comparison with 3% diclofenac gel (Solaraze, medicinal product). It is performed in accordance with both the laws in force for clinical trials with medical devices and those with medicinal products.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years and < 90 years
* Actinic keratosis grade I (mild) or II (moderate) according to the definition by Olsen with palpable or clinically/dermatoscopically apparent keratosis
* Either lesions being well accessible/treatable by the patient or presence of a second person to do the daily applications
* Written informed consent by the patient

Exclusion Criteria:

* Number of initial lesions to be treated ≥ 6
* Overall size of the area to be treated > 25 cm2
* Size (maximum diameter) of single lesion to be treated > 20 mm
* Lesions in close proximity to the eyes, eyelids, nostrils, mouth or mucosal tissue
* Need for topical treatment of cancerous area
* Presence of a relapsing, persistent, indurated, thickened, painful, bleeding, ulcerated and/or rapidly growing lesion
* Existing skin cancer (all forms of skin cancer incl. basal-cell carcinoma and squamous cell carcinoma) in the area to be treated in this study
* Dermal injuries, skin infection or exfoliative dermatitis in the area to be treated in this study
* Other skin diseases in the area to be treated in this study that affect the diagnostic assessment
* Pharmacological or physical local therapy of actinic keratosis (or application of the active ingredients used in the pharmacological therapy) in the area to be treated in this study during the last 4 weeks
* Primary or secondary immunodeficiency
* Treatment with interferons, interferon inducers, immunomodulators or systemic corticosteroids during the last 4 weeks
* Treatment with oral isotretinoin during the last 6 months
* Intracranial bleeding in the medical history or generally increased primary bleeding tendency
* Known intolerance/hypersensitivity to one of the ingredients of the investigational products, especially to diclofenac, parabens or benzyl alcohol as well as to NSAIDs, in particular acetylsalicylic acid
* Pregnancy and lactation
* Women of child-bearing potential either wishing to become pregnant or without effective contraception
* Other serious diseases, which are (according to the investigator's assessment) in conflict with the study participation (i.a. also in view of risk factors for a severe course of a potential COVID-19 disease in case of a SARS-CoV-2 infection)
* Obvious unreliability or lack of cooperation
* Known addiction to alcohol, medicinal products or drugs
* Dependency on the sponsor or an investigator
* Participation in a clinical trial during the last 30 days
* Previous participation in the present clinical trial
* Participation of a family member (in the same household) in the present clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2020-10-14 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Treatment success | At the control visit at the end of treatment ("EOT", i.e. for Solcera/Placebo at the end of cycle 1, 2 or 3 (each cycle is 56 days, number of cycles depends on course of remission), for Solaraze day 60)
  Treatment success, defined as complete, dermatoscopically confirmed remission of all initial actinic keratosis (AK) lesions identified at treatment start that have been treated with the investigational product ("Complete Clearance")

SECONDARY OUTCOMES:
Treatment success | For Solaraze at day 90
  Treatment success, defined as complete, dermatoscopically confirmed remission of all initial AK lesions identified at treatment start that have been treated with the investigational product ("Complete Clearance")
(Healing) status of AK lesions | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  (Healing) status of AK lesions (number of proliferating lesions, unchanged/stable lesions, lesions being in remission or showing partial remission, lesions with complete remission, and relapses; overall and grouped by localisation and size (0-5 mm, 6-10 mm, 11-15 mm, 16-20 mm)); analysed for a) initial AK lesions identified at treatment start that have been treated with the investigational product, b) new AK lesions appearing in the treated area after treatment start, c) all AK lesions (i.e. a) + b))
Overall number of AK lesions | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Overall number of initial AK lesions identified at treatment start that have been treated with the investigational product (i.e. without AK lesions with complete remission)
Mean size of AK lesions | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Mean size of initial AK lesions identified at treatment start that have been treated with the investigational product (lesion size determined by largest diameter)
Treatment success | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Treatment success (complete, dermatoscopically confirmed remission of lesions) analysed for a) initial AK lesions identified at treatment start that have been treated with the investigational product, b) new AK lesions appearing in the treated area after treatment start, c) all AK lesions (i.e. a) + b))
Partial clearance | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Number of patients with "partial clearance" (i.e. all patients with at least 75% of the initial AK lesions identified at treatment start being assessed with "complete remission")
Reduction of AK lesion number | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Reduction of AK lesion number per patient (in % compared to the number of initial AK lesions identified at treatment start) analysed for initial AK lesions identified at treatment start that have been treated with the investigational product
Clinical response | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Clinical response, i.e. the number of patients with at least one AK lesion being assessed with "complete remission"
Lesion-based treatment success (without consideration of relapses) | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Number of initial AK lesions identified at treatment start that have been treated with the investigational product, which showed "complete remission" at least once between treatment start and EOT
Lesion-based treatment success (with consideration of relapses) | At all control/follow-up visits with evaluation of lesions (i.e. for Solcera/Placebo 8 weeks (+ potentially 16 weeks) and 24 weeks after treatment start; for Solaraze Day 30, Day 60, Day 90, 24 weeks)
  Number of initial AK lesions identified at treatment start that have been treated with the investigational product, which showed "complete remission" at the respectively analysed visit
Patients with relapse | Analysed at the follow-up visit 24 weeks after treatment start for the time period between treatment start and the follow-up visit
  Number of patients with at least one initial AK lesion being assessed as "relapse" after previous "Complete Clearance" (definition see above), analysed for the time period between treatment start and the follow-up visit after 24 weeks and analysed in reference to a) the number of all patients and b) the number of those patients with previous "Complete Clearance"
Lesions with relapse | Analysed at the follow-up visit 24 weeks after treatment start for the time period between treatment start and the follow-up visit
  Number of initial AK lesions being assessed as "relapse", analysed for the time period between treatment start and the follow-up visit after 24 weeks and analysed in reference to a) the number of all initial lesions and b) the number of those initial lesions with previous "complete remission"
Efficacy assessment by physician | At EOT (i.e. for Solcera/Placebo at the end of cycle 1, 2 or 3 (each cycle is 56 days, number of cycles depends on course of remission), for Solaraze day 60) and at the follow-up visit 24 weeks after treatment start
  Assessment of the efficacy (scale based on school grades 1-6) by the treating physician
Efficacy assessment by patient | At EOT (i.e. for Solcera/Placebo at the end of cycle 1, 2 or 3 (each cycle is 56 days, number of cycles depends on course of remission), for Solaraze day 60) and at the follow-up visit 24 weeks after treatment start
  Assessment of the efficacy (scale based on school grades 1-6) by the patient
Tolerability assessment by physician | At EOT (i.e. for Solcera/Placebo at the end of cycle 1, 2 or 3 (each cycle is 56 days, number of cycles depends on course of remission), for Solaraze day 60) and at the follow-up visit 24 weeks after treatment start
  Assessment of the tolerability (scale based on school grades 1-6) by the treating physician
Tolerability assessment by patient | At EOT (i.e. for Solcera/Placebo at the end of cycle 1, 2 or 3 (each cycle is 56 days, number of cycles depends on course of remission), for Solaraze day 60) and at the follow-up visit 24 weeks after treatment start
  Assessment of the tolerability (scale based on school grades 1-6) by the patient
Overall assessment by physician | At EOT (i.e. for Solcera/Placebo at the end of cycle 1, 2 or 3 (each cycle is 56 days, number of cycles depends on course of remission), for Solaraze day 60) and at the follow-up visit 24 weeks after treatment start
  Overall assessment (scale based on school grades 1-6) by the treating physician
Overall assessment by patient | At EOT (i.e. for Solcera/Placebo at the end of cycle 1, 2 or 3 (each cycle is 56 days, number of cycles depends on course of remission), for Solaraze day 60) and at the follow-up visit 24 weeks after treatment start
  Overall assessment (scale based on school grades 1-6) by the patient
Adverse Events, Serious Adverse Events, Adverse Reactions | In the time period between start of treatment and the follow-up visit (24 weeks after treatment start)
  Number and frequency of Adverse Events, Serious Adverse Events and Adverse Reactions
Dropouts | In the time period between start of treatment and the follow-up visit (24 weeks after treatment start)
  All dropouts (incl. specification of reason and date)
Compliance | Analysed for the respective time period of scheduled product application, i.e. Day 0 until Day 60 for Solaraze and 1-3x 28 days (depeding on number of cycles) for Solcera/Placebo
  Compliance of the patients with the application schedule of the respective investigational product (based on entries in the patient diary and only overruled by the weight of returned investigational products in case of clear discrepancies)

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Reinhold, Prof., Study Director — MVZ - Dermatologisches Zentrum Bonn GmbH
Locations (18):
- Germany (18):
  - Hautmedizin Bad Soden, Bad Soden
  - MVZ - Dermatologisches Zentrum Bonn GmbH, Bonn
  - Hautzentrum Köln, Cologne
  - Proderma Studienzentrum, Dülmen
  - Hautarztpraxis Falkensee, Falkensee
  - Hautzentrum Südbaden, Freiburg im Breisgau
  - Hautarztzentrum Hamm, Hamm
  - Praxis Dres. Med. Markus Kaspari und Florian Schenk, Hanover
  - Durani Cosmetics GmbH, Heidelberg
  - Hautarztpraxis Ibbenbüren, Ibbenbueren
  - Praxis Dres. K.-H. Vehring/U. Amann, Lingen
  - Zentderma GBR, Mönchengladbach
  - Haut- und Laserzentrum, Potsdam
  - Hautarztpraxis Asefi/Sadjadi, Simmern
  - Hautarztpraxis Leitz und Kollegen, Stuttgart
  - Hautarztpraxis Vilshofen, Vilshofen
  - Centroderm GmbH, Wuppertal
  - Hautzentrum Wuppertal, Wuppertal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinhold U, Leitz N, Dominicus R, Szabo EL, Dirschka T, Popp G, Fischer TC, Adamini N, Ostendorf R, Asefi M, Durani H, Holting T, Amann U, Kreuziger F, Assmann T, Bruning H, Freitag L, Hoffmann K, Gedschold R. KOH 5% solution versus diclofenac 3% for the treatment of actinic keratosis - Results from a three-armed RCT. J Eur Acad Dermatol Venereol. 2025 Sep 25. doi: 10.1111/jdv.70069. Online ahead of print. PMID 40996107